CLINICAL TRIAL: NCT05471830
Title: REal-World Treatment Outcomes of Oral-Anticoagulants Among Patients With Atrial Fibrillation - Patient Survey - RETAF-PS
Brief Title: An Observational Study (Called RETAF-PS) Using a Patient Survey to Learn More About Treatment Outcomes in Patients With Irregular and Often Rapid Heartbeat (Atrial Fibrillation) Treated With Apixaban in a Real World Setting
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22155
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Prevention of Thromboembolic Events; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient survey: Survey-eligible patients with Commercial or Medicare Advantage health insurance who are current/past users of sMRA therapies and diagnosed with chronic kidney disease (CKD), type 2 diabetes (T2D) or heart failure (HF).
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — No drug will be provided to participants. Patients follow routine clinical practice/administration.

SUMMARY:
This is an observational study in which data from people with atrial fibrillation who received or are currently receiving the drug apixaban to prevent thromboembolic events (blood clots that travel through the blood stream to plug another smaller vessel) are studied. In observational studies, only observations are made without specified advice or interventions.

Atrial Fibrillation (AF) is a condition of having irregular and often rapid heartbeat. AF can lead to the formation of blood clots in the heart and to embolism, a condition that happens when a blood clot travels through the blood stream to plug another smaller vessel. This can lead to serious and life-threatening conditions, such as a stroke. A stroke occurs because the brain tissue beyond the blockage no longer receives nutrients and oxygen so that brain cells die. As strokes arising from AF can involve extensive areas of the brain, it is important to prevent them.

Blood clots are formed in a process known as coagulation. This is a complex series of steps that must occur in a specific sequence.

Medications are already available to prevent the formation of blood clots. When taken by mouth (orally), they are known as oral anticoagulants (OACs). OACs decrease the risk of the above-mentioned serious and life-threatening conditions. The main side effect of OACs is an increase of the risk of bleeding.

In the beginning, there was only one main class of OAC called vitamin k antagonists (VKAs) prescribed in usual practice. VKAs work by lowering the number of coagulation factors in the blood. Over the years, newer OAC medications have become available which act more specifically by interrupting one or more of the coagulation steps and preventing the blood from clotting. The study treatment apixaban works by blocking a very specific step in the blood clotting process, the activation of a protein called Factor Xa. Newer OACs are also called direct oral anticoagulants (DOACs). DOACs require less monitoring by doctors, but an increased risk of bleeding remains.

Bleedings can be an important reason for stopping therapy. One type of bleeding called patient relevant bleeding (PRB) has not been intensely studied so far. PRB is a type of minor bleeding which is bothersome, but which does not require medical treatment as it has no important impact on a person's health.

It needs to be distinguished from so called clinically relevant non-major bleeding (CRNMB). CRNMB stands for a type of bleeding which may have an important impact on a person's health and needs medical attention, but when treated, is not likely to have a negative impact on a person's health.

Only limited information is available for PRB and CRNMB related to the treatment with DOACs in real-world settings.

In this study, researchers want to collect more data about how often PRB and CRNMB occur in people with AF treated with apixaban. In addition, researchers want to learn how these medical problems affect the treatment with apixaban under real-world conditions. To do this, researchers will count the number of participants in usual practice

* who have PRB or CRNMB and who are being treated with apixaban at the time of this ongoing study or who have recently taken this drug, but have switched to another OAC,
* who have PRB or CRNMB and have decided to stop or to continue their treatment with apixaban.

In addition, characteristics of each participant and the reason for continuation or discontinuation of apixaban will be collected and described. The data for this study will come from patient surveys.

Besides this data collection, no further tests or examinations are planned in this study.

The participants who take their apixaban treatment during this study will receive their treatments as prescribed by their doctors during routine practice according to the approved product information.

The data will be from participants who will be identified for the survey using last 12-months data from the database called HealthCore Integrated Research Database (HIRD). The data will be collected for each participant for 12 months before the participant starts the survey. The study will end as soon as the planned number of surveys has been reached or at the end date of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Commercial or Medicare Advantage health insurance (both medical and pharmacy benefits) during the patient identification period (most recent 12-months of HIRD claims data at the time the patient sample is identified and extracted).
* Age ≥45 years at the end of the patient identification period.
* At least one medical claim with an ICD-10-CM diagnosis code of AF during the patient identification period.
* At least one pharmacy claim for apixaban during the patient identification period; the date of the most recent pharmacy claim will be the patient sample claims index date.

Exclusion Criteria:

* None

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of survey-eligible, current health plan members with Commercial or Medicare Advantage health insurance who have at least one medical claim with an international classification of disease, 10th revision (ICD-10) diagnosis code for AF and at least one pharmacy claim for apixaban in the HealthCore Integrated Research Database (HIRD). The HIRD will be used as a sampling frame to identify a purposive sample of survey-eligible patients.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation history | Up to 12 months
The occurrence of PRB and CRNMB events and if bleeding was the reason for skipping doses, temporarily pausing, or completely stopping, or changing dose, or switch to other treatment (if occurred) | Up to 12 months
  The questions are designed for participants who are current users of apixaban.
  PRB stands for patient relevant bleeding. CRNMB stands for clinically relevant non-major bleed.
The occurrence of PRB and CRNMB events and if bleeding(s) were reasons for skipped doses, temporarily paused or completely stopped (if occurred) apixaban therapy | Up to 12 months
  The questions are designed for participants who have discontinued apixaban.
Claims-based descriptive analysis of patient demographics characteristics | Up to 12 months
Claims-based descriptive analysis of patient clinical characteristics | Up to 12 months
The occurrence of stroke events during the 12 months prior to the survey date | Up to 12 months

SECONDARY OUTCOMES:
Patient perceptions regarding anticoagulation therapy | Up to 12 months
  Questions for patients who are never on apixaban but current or past use of other anticoagulant questions
Patient perceptions on risk of stroke and bleeding and reasons for not initiated an anticoagulant medication | Up to 12 months
  Questions for participants who were never on anticoagulant treatments
Number of days the participants had apixaban on-hand during the time period between the first prescription within the last 12 months and the survey date (Apixaban adherence) | Up to 12 months
Number of participants who did not have a break in apixaban therapy during the period of time between the first prescription within the last 12-month from the survey date and the survey date (Apixaban persistence) | Up to 12 months
Number of physician office visits during the 12 months prior to the survey date | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.